CLINICAL TRIAL: NCT06304987
Title: The Efficacy and Safety of Preoperative Neoadjuvant Chemoradiation Combined With PD-1 Inhibitor and PCSK9 Inhibitor in the Treatment of pMMR/MSS Locally Advanced Middle and Low Rectal Cancer: a Multicenter Study, Prospective, Randomized Controlled Study
Brief Title: Neoadjuvant Chemoradiotherapy Combined With PD-1 Inhibitor and PCSK9 Inhibitor for pMMR/MSS Locally Advanced Mid-low Rectal Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Beijing Friendship Hospital (Other)
Collaborators: Peking Union Medical College Hospital (Other); Peking University Cancer Hospital & Institute (Other); Changhai Hospital (Other)
Responsible Party: Principal Investigator, Zhongtao Zhang, professor, Beijing Friendship Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BFH-niCRT-05
Record Dates: First submitted 2024-03-05; First posted 2024-03-12 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Locally Advanced Rectal Cancer
Keywords: pMMR/MSS; PD-1; PCSK9; chemoradiation; neoadjuvant
MeSH Terms: interventions — Immune Checkpoint Inhibitors

STUDY DESIGN:
Intervention Model Description: Experimental: Neoadjuvant chemoradiotherapy combined with PD-1 inhibitor and PCSK9 inhibitor Control: Neoadjuvant chemoradiotherapy combined with PD-1 inhibitor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CRT+PD-1 inhibitor+PCSK9 inhibitor (Experimental): Receive long-course radiotherapy in weeks 1-5: 50 Gy/25 f, 2 Gy/day, days 1-5/week; for 5 consecutive weeks; Simultaneously receive 30 days of capetabine treatment at weeks 1-2, weeks 3-5, and weeks 6-8, 825-1000mg/m2, bid, po, days 1-5/week; PD-1 inhibitor: 200mg, iv.gtt, single dose Infusion, a cycle of 21 days, a total of 3 cycles. Carry out at 2 weeks (days 8-14), 5 weeks (days 29-35), and 8 weeks (days 50-56) after the start of radiotherapy; PCSK9 inhibitor: 600 mg, subcutaneous injection, 1, 7 weeks.
  Interventions: Combination Product: Long-course chemoradiation and PD-1 inhibitor, without PCSK9 inhibitor
- CRT+PD-1 inhibitor (Active Comparator): Receive long-course radiotherapy in weeks 1-5: 50 Gy/25 f, 2 Gy/day, days 1-5/week; for 5 consecutive weeks; Simultaneously receive 30 days of capetabine treatment at weeks 1-2, weeks 3-5, and weeks 6-8, 825-1000mg/m2, bid, po, days 1-5/week; PD-1 inhibitor: 200mg, iv.gtt, single dose Infusion, a cycle of 21 days, a total of 3 cycles. Carry out at 2 weeks (days 8-14), 5 weeks (days 29-35), and 8 weeks (days 50-56) after the start of radiotherapy.
  Interventions: Combination Product: Long-course chemoradiation and PD-1 inhibitor, with PCSK9 inhibitor

INTERVENTIONS:
Combination Product: Long-course chemoradiation and PD-1 inhibitor, with PCSK9 inhibitor — In long-course chemoradiotherapy (CRT) + PD-1 inhibitor for LARC patients, the experimental group used concurrent PCSK9 inhibitor, and the active comparison group did not use PCSK9 inhibitor.
  Arms: CRT+PD-1 inhibitor
Combination Product: Long-course chemoradiation and PD-1 inhibitor, without PCSK9 inhibitor — In long-course chemoradiotherapy (CRT) + PD-1 inhibitor for LARC patients, the experimental group used concurrent PCSK9 inhibitor, and the active comparison group did not use PCSK9 inhibitor.
  Arms: CRT+PD-1 inhibitor+PCSK9 inhibitor

SUMMARY:
This is a multicenter, prospective, randomized controlled study to evaluate the effectiveness and safety of neoadjuvant chemoradiotherapy combined with PD-1 inhibitor and PCSK9 inhibitor in the treatment of patients with pMMR/MSS locally advanced middle and low rectal cancer.

DETAILED DESCRIPTION:
This study included patients with locally advanced low rectal cancer as research subjects, and evaluated the efficacy and safety of neoadjuvant chemoradiotherapy combined with PD-1 inhibitor (Sintilimab) and PCSK9 inhibitor (Tafolecimab) or neoadjuvant chemoradiotherapy combined with PD -1 (Sintilimab) for patients with locally advanced rectal cancer. The primary endpoints of the study are clinical complete response (cCR) (including imaging and endoscopic complete response) and pathological complete response (pCR). Secondary endpoints are major pathological response rate (MPR), objective response rate (ORR), disease-free survival (DFS), overall survival (OS), organ preservation rate (OPR), and neoadjuvant rectal (NAR) score, quality of life score (QoL), safety and tolerability.

ELIGIBILITY:
Inclusion Criteria:

1. Sign a written informed consent form and voluntarily join this study;
2. Age 18-75 years old, male or female;
3. Pathologically confirmed adenocarcinoma of the rectum;
4. Clinically staged as II~III stage by MRI (according to the 8th edition of AJCC);
5. Tumor lower edge distance from the anal margin ≤10cm;
6. Able to undergo surgical resection;
7. Able to swallow pills normally;
8. ECOG PS 0-1;
9. No prior anti-tumor therapy for rectal cancer, including radiotherapy, chemotherapy, surgery, etc.;
10. Planning to undergo surgical treatment after completing neoadjuvant therapy;
11. No contraindications for surgery;
12. Normal major organ function, including:

    1. Blood routine examination (no blood or blood products transfusion within 14 days before the first treatment, no use of G-CSF or other hematopoietic stimulating factors for correction):

       * Neutrophil count ≥1.5×109/L
       * Platelet count ≥100×109/L
       * Hemoglobin ≥90 g/L
    2. Blood biochemistry:

       * Total bilirubin ≤1.5×ULN
       * ALT ≤ 2.5×ULN, AST ≤ 2.5×ULN,
       * Serum creatinine ≤1.5×ULN, or creatinine clearance rate ≥50 mL/min (Cocheroft-Gault formula)
    3. Coagulation function:

       * International normalized ratio (INR) ≤ 1.5×ULN
       * Activated partial thromboplastin time (APTT) ≤ 1.5×ULN
       * Female subjects of childbearing potential should have a negative serum pregnancy test within 72 hours before the start of study drug administration, and effective contraception should be used during the trial period and for at least 3 months after the last dose (such as intrauterine devices, contraceptive pills, or condoms); for male subjects with female partners of childbearing potential, effective contraception should be used during the trial period and for 3 months after the last dose.

Exclusion Criteria:

1. History of allergy to monoclonal antibodies, PD-1 monoclonal antibodies, capecitabine, or oxaliplatin;
2. History of receiving or currently receiving any of the following treatments:

   1. Any surgery, radiotherapy, chemotherapy, targeted therapy, immunotherapy, etc., for tumors;
   2. Use of immunosuppressive drugs or systemic steroid therapy to achieve immunosuppression (dose >10mg/day prednisone or equivalent) within 2 weeks before the first use of the study drug; inhalation or local use of steroids and adrenal cortical hormone replacement therapy with a dose >10mg/day prednisone or equivalent is allowed in the absence of active autoimmune diseases;
   3. Receipt of attenuated live vaccines within 4 weeks before the first use of the study drug;
   4. Underwent major surgery or had severe trauma within 4 weeks before the first use of the study drug;
3. Active autoimmune diseases or history of autoimmune diseases, including but not limited to: interstitial pneumonia, enteritis, hepatitis, pituitary inflammation, vasculitis, nephritis, hyperthyroidism, hypothyroidism (considered for inclusion after hormone replacement therapy); psoriasis or childhood asthma/allergies that have completely resolved and do not require any intervention in adulthood may be considered for inclusion, but patients requiring bronchodilators for medical intervention are not eligible for inclusion;
4. History of immunodeficiency, including HIV positive, or acquired or congenital immunodeficiency diseases, or history of organ transplantation or allogeneic bone marrow transplantation;
5. Presence of poorly controlled clinical symptoms or diseases of the heart, including but not limited to: (1) NYHA class II or above heart failure, (2) unstable angina pectoris, (3) myocardial infarction within the past year, (4) clinically significant supraventricular or ventricular arrhythmias that have not been clinically intervened or poorly controlled after clinical intervention;
6. Severe infection (CTCAE > grade 2) within 4 weeks before the first use of the study drug, such as severe pneumonia requiring hospitalization, septicemia, complications of infection, etc.; baseline chest imaging suggests active pulmonary inflammation, presence of symptoms and signs of infection within 14 days before the first use of the study drug or requiring oral or intravenous antibiotic therapy, except for prophylactic use of antibiotics;
7. Active pulmonary tuberculosis infection found through medical history or CT examination, or a history of active pulmonary tuberculosis infection within the past year before enrollment, or a history of active pulmonary tuberculosis infection more than 1 year ago but without proper treatment;
8. Active hepatitis B (HBV DNA ≥ 2000 IU/mL or 104 copies/mL), hepatitis C (HCV antibody positive, and HCV RNA higher than the lower limit of detection of the assay);
9. Diagnosed with other malignant tumors within 5 years before the first use of the study drug, unless they have a low risk of metastasis or death (5-year survival rate > 90%), such as adequately treated basal cell carcinoma or squamous cell skin cancer or carcinoma in situ of the cervix, may be considered for inclusion;
10. Pregnant or lactating women;
11. Judged by the investigator to have other factors that may lead to premature termination of the study, such as having other serious diseases (including mental illnesses) requiring concomitant treatment, alcoholism, drug abuse, family or social factors, factors that may affect the safety or compliance of the subject.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
CR | pCR :within 10 days after surgery;cCR :12-13 weeks after radiotherapy ends
  complete response rate=(number of pathological complete responses + number of clinical complete responses)/total number of patients
AE rate | during treatment
  Adverse event rate

SECONDARY OUTCOMES:
NAR score | within 10 days after surgery
  Neoadjuvant rectal（NAR）score：It is based on the scoring criteria of preoperative treatment
OPR | immediately after surgery
  organ preservation rate
ORR | within 10 days after surgery
  objective response rate
immune-related adverse event rate | up to 30th day after surgery
  adverse event rate that is deemed to be associated with PD-1 inhibition

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Beijing Friendship Hospital, Beijing, Beijing Municipality

IPD SHARING:
Plan to Share IPD: No
Export of individual patient data is a sensitive issue according to current Chinese laws.

REFERENCES:
- [Background] Liu X, Bao X, Hu M, Chang H, Jiao M, Cheng J, Xie L, Huang Q, Li F, Li CY. Inhibition of PCSK9 potentiates immune checkpoint therapy for cancer. Nature. 2020 Dec;588(7839):693-698. doi: 10.1038/s41586-020-2911-7. Epub 2020 Nov 11. PMID 33177715
- [Background] Cohen J, Pertsemlidis A, Kotowski IK, Graham R, Garcia CK, Hobbs HH. Low LDL cholesterol in individuals of African descent resulting from frequent nonsense mutations in PCSK9. Nat Genet. 2005 Feb;37(2):161-5. doi: 10.1038/ng1509. Epub 2005 Jan 16. PMID 15654334
- [Background] Yang Z, Zhang X, Zhang J, Gao J, Bai Z, Deng W, Chen G, An Y, Liu Y, Wei Q, Han J, Li A, Liu G, Sun Y, Kong D, Yao H, Zhang Z. Rationale and design of a prospective, multicenter, phase II clinical trial of safety and efficacy evaluation of long course neoadjuvant chemoradiotherapy plus tislelizumab followed by total mesorectal excision for locally advanced rectal cancer (NCRT-PD1-LARC trial). BMC Cancer. 2022 Apr 27;22(1):462. doi: 10.1186/s12885-022-09554-9. PMID 35477432
- [Background] Abifadel M, Varret M, Rabes JP, Allard D, Ouguerram K, Devillers M, Cruaud C, Benjannet S, Wickham L, Erlich D, Derre A, Villeger L, Farnier M, Beucler I, Bruckert E, Chambaz J, Chanu B, Lecerf JM, Luc G, Moulin P, Weissenbach J, Prat A, Krempf M, Junien C, Seidah NG, Boileau C. Mutations in PCSK9 cause autosomal dominant hypercholesterolemia. Nat Genet. 2003 Jun;34(2):154-6. doi: 10.1038/ng1161. PMID 12730697